CLINICAL TRIAL: NCT02796001
Title: Hallmarks of Protective Immunity in Sequential Rhinovirus Infections in Humans
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Ronald B Turner, Professor of Pediatrics, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 16-0055
Record Dates: First submitted 2016-06-07; First posted 2016-06-10 (Estimated); Results first posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — viral protein 1, rhinovirus

STUDY DESIGN:
Intervention Model Description: Volunteers who were infected with RV16 by experimental challenge were eligible for participation by re-challenge with either RV16 or RV39 to assess the host response to homologous or heterologous rechallenge.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- RV16 infected volunteers re-challenged with RV16 (Active Comparator): volunteers re-challenged with RV16
  Interventions: Biological: human rhinovirus
- RV infected volunteers re-challenged with RV39 (Active Comparator): volunteers re-challenged with RV39
  Interventions: Biological: human rhinovirus
- RV infected not rechallenged (Other): Volunteers who were infected with RV16 and eligible for re-challenge but who were not re-challenged due to voluntary withdrawal (3) or removal for exclusion criteria
  Interventions: Other: no intervention

INTERVENTIONS:
Biological: human rhinovirus — human rhinovirus
  Arms: RV infected volunteers re-challenged with RV39; RV16 infected volunteers re-challenged with RV16
Other: no intervention — 4 volunteers were not re-challenged and did not participate in the second challenge
  Arms: RV infected not rechallenged

SUMMARY:
The primary objective of this study is to assess the relationship between rhinovirus specific T-cell immunity and the human host response to primary rhinovirus challenge and subsequent secondary challenge with either homologous or heterologous rhinovirus serotypes.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the relationship between RV-specific T-cell immunity and the human host response to primary RV challenge and subsequent secondary challenge with either homologous or heterologous RV serotypes. The overall hypothesis that will be addressed by the mechanistic studies in this proposal is that T helper (Th) and T follicular helper (Tfh) cells directed against conserved RV epitopes expand upon RV exposure and some of these cells persist as stable cross-reactive memory populations capable of displaying lineage-specific protective functions upon re-infection with related or unrelated strains of RV. The human specimens collected in this study will be analyzed with a variety of state-of-the-art techniques to provide an in depth description of T-cell responses to RV infection, and the correlation of these responses with viral infection, antibody responses, and illness. Beyond this objective, by using a systems biology approach, we aim to gain new insight into the role of diverse cell types involved in adaptive immunity to RV. .

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 18-40 years of age
2. Subject must read and sign a copy of the approved Consent Form
3. Subject must have a serum neutralizing antibody titer of ≤1:2 to rhinovirus type 39 and rhinovirus type 16
4. Female subjects must be using an effective birth control method.
5. Total IgE <150 IU/ml.

Exclusion Criteria:

1. Any clinically significant abnormalities of the upper respiratory tract
2. Any clinically significant acute or chronic respiratory illness
3. Any clinically significant bleeding tendency by history
4. Hypertension that requires treatment with antihypertensive medications
5. History of angina or other clinically significant cardiac disease
6. Any upper respiratory infection or allergic rhinitis in the two weeks prior to the start of the study
7. Any medical condition that in the opinion of the Investigator is cause for exclusion from the study
8. Use of any anti-inflammatory (steroids or NSAIDs) or cough/cold preparation in the 1 month prior to the study
9. Regular use of tobacco in the last 6 months (ie. more than 2 days out of 7) or inability to refrain from smoking during the study
10. Inability to refrain from the use of common cold therapies in the 5 days after each rhinovirus challenge.
11. Participation in any other clinical drug trial in the month prior to the study
12. Female subjects with a positive urine pregnancy screen.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Turner, MD, Principal Investigator — Univ of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Barone SM, Paul AG, Muehling LM, Lannigan JA, Kwok WW, Turner RB, Woodfolk JA, Irish JM. Unsupervised machine learning reveals key immune cell subsets in COVID-19, rhinovirus infection, and cancer therapy. Elife. 2021 Aug 5;10:e64653. doi: 10.7554/eLife.64653. PMID 34350827

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteers who participated in the study were individuals who had previously been challenged and infected with RV16 in the human rhinovirus experimental challenge model and agreed to be re-challenged with either RV16 or RV39
Pre-assignment Details: Volunteers were initially challenged with RV16 to provide a uniform baseline for the subsequent randomization and re-challenge with either a homologous serotype (RV16) or a heterologous serotype (RV39). 46 subjects met the baseline criteria but 3 declined further participation and 1 was ill on the day of re-challenge and was removed from the study by the investigator. 42 subjects were randomized and re-challenged with rhinovirus.
Groups:
- RV16 Infected Volunteers Re-challenged With RV39: volunteers re-challenged with RV39
  human rhinovirus: human rhinovirus
- no Intervention: 4 volunteers were infected with RV16 and were eligible to be randomized to re-challenge. Three of these volunteers declined re-challenge and one was removed from the study prior to re-challenge
Period: Overall Study
Arm/Group | RV16 Infected Volunteers Re-challenged With RV16 | RV16 Infected Volunteers Re-challenged With RV39 | no Intervention
Started | 20 | 22 | 4
Completed | 20 | 22 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Volunteers re-challenged with RV16 or RV39
Groups:
- no Intervention: 4 volunteers were infected with RV16 and were eligible for re-challenge. Three volunteers declined re-challenge and one was removed from the study prior to re-challenge
- Total: Total of all reporting groups
Arm/Group | RV16 Infected Volunteers Re-challenged With RV16 | RV16 Infected Volunteers Re-challenged With RV39 | no Intervention | Total
Number analyzed (Participants) | 20 | 22 | 4 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.7 (2.43) | 19.8 (1.87) | 19.25 (0.5) | 20.1 (1.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 2 | 24
  Male | 8 | 12 | 2 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 15 | 19 | 3 | 37
  More than one race | 2 | 0 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 22 | 4 | 46
previously infected with RV16 [Count of Participants; unit: Participants] | 20 | 22 | 4 | 46

OUTCOME MEASURES:

1. Primary Outcome: Virus Infection
Description: Number infected after re-challenge with RV16 compared to RV39 as determined by virus isolation in cell culture or viral serology
Time Frame: Volunteers were cultured daily for detection of virus shedding for 5 days after the virus re-challenge and serum was collected for viral serology 4 weeks after virus re-challenge
Population: all volunteers re-challenged
Measure: Count of Participants; unit: Participants
Arm/Group | RV16 Infected Volunteers Re-challenged With RV16 | RV16 Infected Volunteers Re-challenged With RV39
Number analyzed (Participants) | 20 | 22
Participants | 8 | 18

ADVERSE EVENTS:
Time Frame: Adverse events were collected at each study visit from the virus challenge/re-challenge to 15 weeks.
Description: Adverse events were collected by interactive interview with study staff at each study visit between challenge/re-challenge and week 15. 46 subjects were initially challenged with RV16. 42 subjects were re-challenged with either RV16 or RV39. Three subjects voluntarily withdrew from the study before re-challenge and one subject had common cold symptoms on the scheduled day of the re-challenge and was removed from the study by the investigator.
Groups:
- Volunteers Initially Challenged With RV16: Volunteers challenged with RV16 to produce RV16 infected volunteers for subsequent arms
  Human rhinovirus
Arm/Group | Volunteers Initially Challenged With RV16 | RV16 Infected Volunteers Re-challenged With RV16 | RV16 Infected Volunteers Re-challenged With RV39
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/20 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/20 | 0/22
Other Adverse Events (participants affected / at risk) | 2/46 | 1/20 | 1/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Volunteers Initially Challenged With RV16 (N=46) | RV16 Infected Volunteers Re-challenged With RV16 (N=20) | RV16 Infected Volunteers Re-challenged With RV39 (N=22)
bloody nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — increased headache after day 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT02796001/Prot_SAP_000.pdf